CLINICAL TRIAL: NCT06246500
Title: Severe Head Trauma: Coagulation and CT-Scan Aggravation.
Acronym: TCA-COAG
Status: Terminated | Type: Observational
Why Stopped: Recruitment issue
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 18-43
Record Dates: First submitted 2021-03-02; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2022-07

CONDITIONS: Head Trauma
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Retrospective, multicenter cohort study describing the biological, radiological and clinical criteria of patients managed for isolated severe head trauma between January 2016 and December 2018.

DETAILED DESCRIPTION:
The objective of the study is to describe the evolution of CTscan lesions in patients with isolated Head Trauma between admission and re-evaluation after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patients informed and did not object to the collection of their medical data for the study
* Patient admitted in Trauma center between January 2016 and December 2018 severe head injury defined by a Glasgow Coma Scale (GCS) < 9 AND/OR Abnormalities on the first brain CT-scan with pathological transcranial Doppler (Vd < 25 cm/s and IP > 1.25)

Exclusion Criteria:

* Abbreviated Injury Score (AIS) head and neck ≤ 3 AND/OR AIS out of head and neck > 3
* Taking drugs that interfere with hemostasis, such as anticoagulant or antiplatelet antiaggregants in preventive or curative doses;
* Patients under guardianship
* Patients still alive at the time of data collection AND opposed to the collection of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient data will be selected retrospectively and consecutively according to in and exclusion criteria. All patient admitted in emergency room between January 2016 and December 2018 severe head injury defined
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Describe the evolution of CT scan lesions between admission and reassessment CT scan | 24 hours
  Number of patient with an aggravation of lesions on CT scan

SECONDARY OUTCOMES:
Mortality | Day 28
  Mortality rate
Causes of death | Day 28
  Causes of death
Describe the coagulation status on admission with severe head trauma trauma | 24 hours
  Fibrinogen level values
Describe the coagulation status on admission with severe head trauma trauma | 24 hours
  Platelet count values
Describe the coagulation status on admission with severe head trauma trauma | 24 hours
  INR values
Describe the coagulation status on admission with severe head trauma trauma | 24 hours
  ROTEM values

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Annecy Genevois, Pringy, France